CLINICAL TRIAL: NCT02641808
Title: Does Follicular Flushing Improve the Outcome in Monofollicular IVF Therapy?
Acronym: Flushing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Principal Investigator, Alexandra Kohl Schwartz, Dr. med., Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-00150
Record Dates: First submitted 2015-12-12; First posted 2015-12-29 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- follicular flushing group (Experimental): Monofollicular IVF therapy with follicular flushing up to five times after aspiration of the follicule at the time to the oocyte pick-up
  Interventions: Other: follicular flushing
- aspiration group (Active Comparator): Monofollicular IVF therapy with aspiration only at the time of the oozyte pick-up
  Interventions: Other: no follicular flushing

INTERVENTIONS:
Other: follicular flushing — Depending on randomisation the follicle is not flushed (group A) or flushed adapted to follicule size (16mm 2ml, 18mm 3ml, and 20mm 4ml etc.) up to five times with (e.g.flushing media with heparin (SynVitro® Flush, Origio, Berlin, Germany). The flushings are collected each in a separate collecting tube (group B). The analysis of the collected oocytes is performed in the IVF lab.
  Arms: follicular flushing group
Other: no follicular flushing
  Arms: aspiration group

SUMMARY:
Follicular aspiration as well as follicular flushing are standardized techniques and have been practiced in polyfollicular IVF (in vitro fertilization) therapy for years. Monofollicular IVF therapy is a standard technique as well. IVF can be done in natural cycles or with a minimal stimulation with clomifen citrate to achieve a monofollicular response. Our study aims to compare follicular aspiration and follicular flushing in monofollicular stimulation. First the investigators want to answer the question whether flushing is beneficial for the oocyte yield. In case of a positive result the investigators want to establish a recommendation about the optimal number of flushings taking into account the duration of the procedure and the pain during manipulation.

DETAILED DESCRIPTION:
There is an increase in mono- and oligofollicular IVF therapies worldwide. With the increase in oligo- and monofollicular IVF techniques, a re-evaluation of the aspiration techniques is necessary. The lower the number of mature follicules, the higher the need to obtain the oocyte. The number of embryos obtained is dependent on the number of oocytes retrieved (Wood 2000).

Von Wolff et al. showed (2013) that, three flushings almost doubled not only the number of aspirated oocytes but also the transfer rate in monofollicular IVF. Oocytes, collected by flushing, were as mature and fertilizable as those aspirated without flushing. Mendez Lozano et al. performed an aspiration without flushing in 79 women and with triple flushing in 47 women. They were stimulated with HMG (human menopausal gonadotropin) and controlled with GnRH (Gonadotropin releasing hormone) antagonists in a semi natural cycle IVF. The percentage of patients with a good embryo was 28.8% in the group without flushing and 37.8% in the group with flushing; however, the difference was not significant. Women with an indication for an IVF therapy and the wish of natural cycle IVF are randomized to the intervention (flushing) or control arm (no flushing). In natural cycle IVF, there is no gonadotropin stimulation. Clomifen citrate (25mg e.g. Serophene®, Merck Serono, from the 6th day of cycle) or singles doses of GnRH-antagonists (e.g. Orgalutran®, MSD, Merck Sharp & Dohme AG) are only given to avoid premature ovulation. Once maturity of the follicle is achieved (follicle size ≥16mm), 5000IU urinary human chorionic gonadotropin (uHCG) is used to trigger ovulation. Oocyte pickup (OPU) is performed 36.5 (36-37) hours after ovulation induction. No anesthesia is used for this procedure. For the aspiration 19 gauge single lumen needles are used. After the aspiration the needle is removed and flushed. Depending on randomisation the follicle is not flushed (group A) or flushed adapted to follicule size (16mm 2ml, 18mm 3ml, and 20mm 4ml etc.) up to five times with (e.g.flushing media with heparin (SynVitro® Flush, Origio, Berlin, Germany). In case more than 1 follicle develops, only the largest follicle is analysed. The flushings are collected each in a separate collecting tube (group B). The analysis of the collected oocytes is performed in the IVF lab. The aspirated fluid is analyzed in the IVF lab by the independent biologist. Pain is monitored by VAS (visual analogue scale) score and time of intervention is measured. In the IVF lab the oocytes are fertilised by ICSI (intracytoplasmatic sperm injection) and the embryo transferred 2-3 days later.

ELIGIBILITY:
Inclusion Criteria:

* Indication for in vitro Fertilisation
* Desire of natural cycle IVF and ICSI fertilisation
* Regular menstrual cycle, both ovaries can be reached for follicule aspiration
* 18-42 years
* size of the follicle ≥16mm
* max. 2 previous embryo transfers

Exclusion Criteria:

* <18 and >42 years
* Preterm ovulation
* >= 3 previous embryo transfers

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Proportion of mature oocytes retrieved | day of intervention

SECONDARY OUTCOMES:
Number of flushings necessary to retrieve the oocyte (intervention arm only) | day of intervention
Fertilisation rate | one day after intervention
Embryo quality (BLEFCO and ASEBIR score) on day 2 after fertilisation | two days after intervention
Transfer rate | 2-3 days after intervention
Pregnancy rate | up to 9 months after the intervention
Pain during intervention measured on a VAS scale | day of intervention
Time used for intervention | day of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra S Kohl Schwartz, MD, Principal Investigator — Reproductive Endocrinologist

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kohl Schwartz AS, Calzaferri I, Roumet M, Limacher A, Fink A, Wueest A, Weidlinger S, Mitter VR, Leeners B, Von Wolff M. Follicular flushing leads to higher oocyte yield in monofollicular IVF: a randomized controlled trial. Hum Reprod. 2020 Oct 1;35(10):2253-2261. doi: 10.1093/humrep/deaa165. PMID 32856073